CLINICAL TRIAL: NCT05089903
Title: Breast Cancer Outreach Among Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Shivan Mehta, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: UPCC 15121; 849863 (Other: UPenn IRB)
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: Mammography; Preventive Screening; Population Health
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- No Order (Experimental)
  Interventions: Behavioral: No Bulk Order
- No Order + Text (NO+T) (Experimental)
  Interventions: Behavioral: Texting; Behavioral: No Bulk Order
- Bulk Order (BO) (Experimental)
  Interventions: Behavioral: Bulk Order
- Bulk Order + Text (BO+T) (Experimental)
  Interventions: Behavioral: Bulk Order; Behavioral: Texting
- Clinician Endorsement (CE) (Experimental)
  Interventions: Behavioral: Clinician Endorsement
- Clinician Endorsement + Text (CE+T) (Experimental)
  Interventions: Behavioral: Texting; Behavioral: Clinician Endorsement
- Standard Messaging (SM) (Experimental)
  Interventions: Behavioral: Standard Endorsement
- Standard Messaging (SM+T) (Experimental)
  Interventions: Behavioral: Texting; Behavioral: Standard Endorsement

INTERVENTIONS:
Behavioral: Bulk Order — A mammogram order will be placed using bulk order technology in the EHR in advance of outreach for all patients.
  Arms: Bulk Order (BO); Bulk Order + Text (BO+T)
Behavioral: Texting — In addition to outreach, patients will receive text messaging with information regarding the importance of screening, how to schedule a mammogram, and locations available for mammography.
  Arms: Bulk Order + Text (BO+T); Clinician Endorsement + Text (CE+T); No Order + Text (NO+T); Standard Messaging (SM+T)
Behavioral: Clinician Endorsement — Outreach informing patients that they are overdue for a mammogram will be signed by the patient's primary care provider.
  Arms: Clinician Endorsement (CE); Clinician Endorsement + Text (CE+T)
Behavioral: No Bulk Order — The outreach will ask patients to contact their PCP's office in order to have a mammogram order placed on their behalf.
  Arms: No Order; No Order + Text (NO+T)
Behavioral: Standard Endorsement — Patient's will receive outreach from the practice informing them that they are overdue for a mammogram.
  Arms: Standard Messaging (SM); Standard Messaging (SM+T)

SUMMARY:
This project aims to evaluate different approaches to increase breast cancer screening among primary care patients at Penn Medicine through a centralized screening outreach program. In a pragmatic trial, the investigators will evaluate different approaches to increase completion of screening among eligible patients, including ordering mammograms in bulk prior to outreach, sending personalized text reminders, and endorsing of the communication by the primary care provider.

DETAILED DESCRIPTION:
While mammograms are recommended by guidelines for early detection of breast cancer, mammogram rates are significantly lower now than they were prior to the initial COVID-19 pandemic surge in early 2020. In this project, the investigators will evaluate different ways of reaching out to eligible patients to encourage them to participate in breast cancer screening. Through letters, texting, and the electronic health record portal (MyPennMedicine (MPM)), the investigators will compare mammogram bulk orders, text messaging, and primary care provider endorsement to traditional outreach messaging with the goal of increasing breast cancer screening uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 40-74
2. Followed by Primary Care with a Penn Medicine PCP listed and at least one visit in the last 2 years
3. Health Maintenance due (default biannual screening starting at age 50 or edit modifier based on input by clinician)

Exclusion Criteria:

1. Currently scheduled for a mammogram
2. History of bilateral mastectomy

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24680 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Mammogram Completion in 3 months | 3 months
  Percent of patients that complete a mammogram

SECONDARY OUTCOMES:
Mammogram Completion in 6 months | 6 months
  Percent of patients that complete a mammogram

OTHER OUTCOMES:
Mammogram Positivity Rate | 3 months
  Percent of mammograms that have positive results
Mammogram Completion by Age Groups | 3 months
  Percent of patients that complete a mammogram by age groups
Mammogram Completion by Race/Ethnicity | 3 months
  Percent of patients that complete a mammogram by race/ethnicity
Mammogram Completion by Insurance Type | 3 months
  Percent of patients that complete a mammogram by insurance type
Mammogram Completion by Median Household Income by Zip Code | 3 months
  Percent of patients that complete a mammogram by Median Household Income by zip code
Positive Mammograms Resulting in Subsequent Care | 3 months
  Percent of patients with a positive mammogram that receive subsequent care
Mammogram Completion by Electronic Patient Portal Status | 3 months
  Percent of patients that complete a mammogram by electronic patient portal status

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Rhodes C, Linn KA, Reitz C, McDonald C, Okorie E, Williams K, Resnick D, Arostegui A, McAuliffe T, Wollack C, Snider CK, Peifer MK, Weinstein SP. Behavioral Interventions to Improve Breast Cancer Screening Outreach: Two Randomized Clinical Trials. JAMA Intern Med. 2024 Jul 1;184(7):761-768. doi: 10.1001/jamainternmed.2024.0495. PMID 38709509